CLINICAL TRIAL: NCT05662033
Title: A Blinded, Randomised, Placebo-controlled Study to Investigate the Safety, Tolerability, and Pharmacokinetics of an Oral Suspension of AZD6793 Following Single and Multiple Ascending Doses in Healthy Subjects, an Open-label Study to Assess the Relative Bioavailability and Food Effect of a Tablet Formulation of AZD6793 in Healthy Subjects and a Blinded, Randomised, Placebo-controlled Study to Investigate the Safety, Tolerability, and Pharmacokinetics of a Tablet Formulation of AZD6793 in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics (PK) of Oral AZD6793 in Healthy and Chronic Obstructive Pulmonary Disease Participants, to Assess the Relative Oral Bioavailability Between Two Formulations, and the Food Effect on the PK of AZD6793 Compared to Fasting State.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: D7860C00001; 2022-002951-21 (EudraCT Number)
Record Dates: First submitted 2022-11-16; First posted 2022-12-22 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Inflammatory Diseases
Keywords: IRAK4 kinase inhibitor; AZD6793

STUDY DESIGN:
Intervention Model Description: The study consists of 4 parts:
  Part 1 (SAD): In this part, healthy participants will be randomised in 5 cohorts (may add up to 3 additional cohorts) to receive AZD6793 with 8 evaluable participants in each cohort.
  Part 2 (MAD): In this part, healthy participants will be randomised in 3 cohorts (may add up to 3 additional cohorts) to receive AZD6793 with 8 evaluable participants in each cohort.
  Part 3 (Bioavailability and Food Effect Cohort): In this cohort, 15 healthy participants will be randomised to receive AZD6793 with 12 evaluable participants.
  Part 4 (COPD Cohort): 15 COPD participants will be randomised in the ratio 2:1 to receive AZD6793 or placebo.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Part 1 (SAD): Cohort 1 (Experimental): 6 Healthy participants will receive a single oral dose A of AZD6793 and 2 healthy participants will receive placebo
  Interventions: Drug: AZD6793; Drug: Placebo
- Part 1 (SAD): Cohort 2 (Experimental): 6 Healthy participants will receive a single oral dose B of AZD6793 and 2 healthy participants will receive placebo
  Interventions: Drug: AZD6793; Drug: Placebo
- Part 1 (SAD): Cohort 3 (Experimental): 6 Healthy participants will receive a single oral dose C of AZD6793 and 2 healthy participants will receive placebo
  Interventions: Drug: AZD6793; Drug: Placebo
- Part 1 (SAD): Cohort 4 (Experimental): 6 Healthy participants will receive a single oral dose D of AZD6793 and 2 healthy participants will receive placebo
  Interventions: Drug: AZD6793; Drug: Placebo
- Part 1 (SAD): Cohort 5 (Experimental): 6 Healthy participants will receive a single oral dose E of AZD6793 and 2 healthy participants will receive placebo
  Interventions: Drug: AZD6793; Drug: Placebo
- Part 2 (MAD): Cohort 1 (Experimental): 6 Healthy participants will receive dose W of AZD6793 and 2 healthy participants will receive placebo once daily on Day 1 and 8 and twice daily on Day 3 to Day 7
  Interventions: Drug: AZD6793; Drug: Placebo
- Part 2 (MAD): Cohort 2 (Experimental): 6 Healthy participants will receive dose X of AZD6793 and 2 healthy participants will receive placebo once daily on Day 1 and 8 and twice daily on Day 3 to Day 7
  Interventions: Drug: AZD6793; Drug: Placebo
- Part 2 (MAD): Cohort 3 (Experimental): 6 Healthy participants will receive dose Y of AZD6793 and 2 healthy participants will receive placebo once daily on Day 1 and 8 and twice daily on Day 3 to Day 7
  Interventions: Drug: AZD6793; Drug: Placebo
- Part 2 (MAD) : Cohort 4 (Experimental): 6 Healthy participants will receive dose Z of AZD6793 and 2 healthy participants will receive placebo once daily on Day 1 and 8 and twice daily on Day 3 to Day 7
  Interventions: Drug: AZD6793; Drug: Placebo
- Part 3: Treatment sequence 1 (Experimental): Participants will receive a single oral dose of test formulation AZD6793 in fasted state, test formulation AZD6793 in fed state following reference formulation AZD6793 in fasted state once on Day 1 of each treatment period.
  Interventions: Drug: AZD6793
- Part 3: Treatment sequence 2 (Experimental): Participants will receive a single oral dose of test formulation AZD6793 in fed state, reference formulation AZD6793 in fasted state following test formulation AZD6793 in fasted state once on Day 1 of each treatment period.
  Interventions: Drug: AZD6793
- Part 3: Treatment sequence 3 (Experimental): Participants will receive a single oral dose of reference formulation AZD6793 in fasted state, test formulation AZD6793 in fasted state following test formulation AZD6793 in fed state once on Day 1 of each treatment period.
  Interventions: Drug: AZD6793
- Part 4 (COPD): Cohort 1 (Experimental): 10 participants with COPD will receive AZD6793 once daily and 5 participants with COPD will receive placebo
  Interventions: Drug: AZD6793; Drug: Placebo

INTERVENTIONS:
Drug: AZD6793 — AZD6793 will be administered orally
Drug: Placebo — Placebo will be administered orally
  Arms: Part 1 (SAD): Cohort 1; Part 1 (SAD): Cohort 2; Part 1 (SAD): Cohort 3; Part 1 (SAD): Cohort 4; Part 1 (SAD): Cohort 5; Part 2 (MAD) : Cohort 4; Part 2 (MAD): Cohort 1; Part 2 (MAD): Cohort 2; Part 2 (MAD): Cohort 3; Part 4 (COPD): Cohort 1

SUMMARY:
The purpose of the study is to assess the safety and tolerability of AZD6793 suspension following oral administration of Single Ascending Dose (SAD) [Part 1] and Multiple Ascending Dose (MAD) [Part 2] in healthy participants.

Additionally, the study will include Part 3 (bioavailability and food effect cohort) to assess the relative oral bioavailability between test formulation and oral suspension (reference formulation) as well as the effect of a high fat high calorie (HFHC) meal on the PK of AZD6793 test formulation, in comparison to fasting conditions, after a single oral dose of AZD6793 in healthy participants.

Part 4 of the study (Chronic Obstructive Pulmonary Disease [COPD] cohort) is intended to evaluate AZD6793 safety, tolerability, and PK profile for the first time in participants with moderate to severe COPD.

Part 1 (SAD), Part 2 (MAD) and Part 3 (Bioavailability and food effect cohort) have been completed. Although it was planned that 5 cohorts would be included in Part 1, only 4 cohorts (32 participants) were included. Part 3 of the study was concluded with 13 healthy participants.

DETAILED DESCRIPTION:
Parts 1, 2, and 3 were conducted in a single center and Part 4 is conducted in 2 centers.

Part 1 of the study will comprise:

* A Screening Period of maximum 28 days (Day -29 to Day -2)
* A Treatment Period during which participants will be resident at the Clinical Unit from Day -1 (the day before IMP administration [Day 1]) until at least 72 hours after IMP administration. Participants will then be discharged on Day 4 if in good health and after all samples have been collected. Depending on the emerging data, the length of the stay at the Clinical Unit may be changed.
* A Follow-up Visit within 6 ± 1 days after the IMP dose (this visit may be done later if indicated, for example, if emerging PK data indicates a longer AZD6793 half-life than was predicted).

Part 2 of the study will comprise:

* A Screening Period of maximum 28 days (Day -29 to Day -2).
* A Treatment Period during which participants will be resident at the Clinical Unit from Day -1 (the day before first IMP administration [Day 1]) until Day 10. participants will receive a single dose of IMP in the morning on Day 1. After a washout of at least 48 hours (depending on PK data from Part 1), participants will be dosed twice daily (12 hours apart) from Day 3 through Day 7. Participants will receive the last dose of IMP in the morning of Day 8. Participants will then be discharged on Day 10 if in good health and after all samples have been collected.
* A Follow-up Visit within 6 ± 1 days after the last IMP dose (this visit may be done later if indicated, for example, if emerging PK data indicates a longer AZD6793 half-life than was predicted).

Part 3 of the study will comprise:

* A Screening Period of maximum 28 days (Day -29 to Day -2).
* A Treatment Period during which participants will be resident at the Clinical Unit from Day -1 until Day 3. Participants will be randomised on Day 1 of Visit 3 to one of 3 treatment sequences and will receive AZD6793 on Day 1 of each treatment period. Dose administration will be separated by a washout period of at least 3 days from the previous IMP dose of each treatment period.
* A Follow-up Visit within 6 ± 1 days after the last IMP dose

Part 4 of the study will comprise:

* A Screening Period of maximum 35 days (Day -35 to -2)
* A Treatment Period of up to 28 days (at least 26 days) of dosing with AZD6793 or placebo. The participants will be admitted to the Clinical Unit on Day -1 and will receive single dose of AZD6793 or placebo on Day 1 and discharged from the Clinical Unit in the evening on Day 1 (12 hours post-dose).
* A Follow--up Visit 6 ± 2 days after the last IMP dose

ELIGIBILITY:
Main Inclusion Criteria:

Parts 1,2 and 3:

* Healthy male or female participants aged 18 to 55 years with suitable veins for cannulation or repeated venepuncture
* Females must have a negative pregnancy test must not be lactating and must be either (a) non-childbearing potential, confirmed by post-menopausal defined as amenorrhea for at least 12 months; documentation of irreversible surgical sterilisation or (b) childbearing potential, i.e., fertile, following menarche and until becoming post-menopausal unless permanently sterile (Must agree to use, with their partner, an approved method of highly effective contraception).
* Male participants and their female partners of childbearing potential must be willing to use highly effective contraception measures and male participants must refrain from donating sperm or fathering a child from the first day of dosing until 3 months after the last dose of IMP.
* Have a BMI between 18 and 30 kg/m2 inclusive and weigh at least 50 kg, at the Screening Visit.

Part 4:

* Male and/or female participants, who have moderate to severe COPD, and aged 40 through 80 years inclusive.
* BMI between 18 to 44.9 kg/m2 at Screening
* Documented history of COPD with a post-bronchodilator FEV1/FVC <0.70 and a post-bronchodilator FEV1 ≥ 30% and < 80% predicted at Screening
* Documented stable inhaled treatment regimen of dual therapy or triple therapy for ≥ 3 months prior to Screening.
* Clinically stable and free from an Acute exacerbation of chronic obstructive pulmonary disease (AECOPD) in the opinion of the Investigator for at least 35 days prior to Day 1
* Females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit, must not be lactating and must be of :

  1. Non-childbearing potential confirmed at screening
  2. If considered of childbearing potential, must agree to use with their partner an approved method of highly effective contraception.
* Male participants and their female partners of childbearing potential must be willing to use highly effective contraception measures and must refrain from donating sperm or fathering a child from first day of dosing until 3 months after last IMP dose.

Main Exclusion Criteria:

Parts 1,2 and 3:

* History or presence of gastrointestinal, hepatic, renal, pancreatic disease or acute disease in these organs.
* History of chronic haematologic disease.
* Diagnosis or history of immunodeficiency or increased susceptibility to severe infection, or a clinically significant infection
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
* Positive or indeterminate QuantiFERON® Tuberculosis (TB) test at screening.
* Any clinically important abnormalities in clinical chemistry, haematology or urinalysis results
* Any positive result on Screening for serum Hepatitis B surface antigen (HBsAg), hepatitis C antibody and Human immunodeficiency virus (HIV).
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting Electrocardiogram (ECG) and any clinically important abnormalities in the 12 lead ECG.
* Known or suspected history of alcohol and drug abuse in the last year.
* Current smokers or those who have smoked or used nicotine products (including e cigarettes) within the previous 3 months.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to AZD6793.
* Excessive intake of caffeine containing drinks or food
* Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
* Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, mega dose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half life
* Plasma donation within one month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to the Screening Visit.
* Parts 2 and 3 only: Participants who have previously received AZD6793.

Part 4:

* Concurrent enrolment in another clinical study involving an investigational treatment
* Participants unable to perform reproducible spirometry according to American Thoracic Society/ European Respiratory Society [ATS/ERS] criteria at Screening
* Any active medical condition or other reason (at Screening, Day -1, and pre-dose) that would interfere with evaluation of the investigational product or interpretation of participant safety or study results, any other clinically relevant abnormal findings on physical examination or laboratory testing at Screening
* Positive or indeterminate QuantiFERON® TB test at Screening. Indeterminate results may be repeated during Screening.
* Major surgery within 8 weeks prior to Screening
* Donation of blood or blood products in excess of 500 mL within 3 months prior to Screening
* History or current diagnosis of cancer, history of an underlying condition that predisposes the participant to infections, known history of severe reaction to any medication, history of allogeneic bone marrow transplant and history of viral, bacterial or fungal infections within 4 weeks prior to randomisation
* Receiving any immunotherapy or immunosuppressive therapy other than corticosteroids within 6 months of randomisation
* Participants taking metformin during Screening or at any time during the study
* Any participant with active hepatitis or Human immunodeficiency virus (HIV)
* History or presence of vitiligo or significant (in the opinion of the Investigator) skin depigmentation for any cause including drugs
* History of clinically significant chronic/active haematology disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Part 1 (SAD): Number of participants with adverse events | From screening up to Follow up visit (Day 6±1)
  Safety and tolerability of AZD6793 following oral administration of SAD in healthy participants.
Part 2 (MAD): Number of participants with adverse events | From screening up to Follow up visit (Day 14±1)
  Safety and tolerability of AZD6793 following oral administration of MAD in healthy participants.
Part 1 (SAD): Number of participants with abnormal findings in vital signs (supine Blood Pressure (BP), pulse, respiratory rate, peripheral oxygen saturation (SpO2) and oral body temperature) | From screening, Treatment Day 1 to Day 4 up to Follow up visit (Day 6±1)
  Safety and tolerability of AZD6793 following oral administration of SAD in healthy participants.
Part 2 (MAD): Number of participants with abnormal findings in vital signs (supine Blood Pressure (BP), pulse, respiratory rate, peripheral oxygen saturation (SpO2) and oral body temperature) | From screening, Treatment Day -1 to Day 10 up to Follow up visit (Day 14±1)
  Safety and tolerability of AZD6793 following oral administration of MAD in healthy participants.
Part 1 (SAD): Number of participants with abnormal findings in 12 Lead electrocardiogram (ECG) | From screening, Treatment Day -1 to Day 4 up to Follow up visit (Day 6±1)
  Safety and tolerability of AZD6793 following oral administration of SAD in healthy participants.
Part 2 (MAD): Number of participants with abnormal findings in 12 Lead electrocardiogram (ECG) | From screening, Treatment Day -1 to Day 10 up to Follow up visit (Day 14±1)
  Safety and tolerability of AZD6793 following oral administration of MAD in healthy participants.
Part 1 (SAD): Number of participants with abnormal findings in 12 Lead Digital electrocardiogram (dECG) | Day 1 to Day 3
  Safety and tolerability of AZD6793 following oral administration of SAD in healthy participants.
Part 2 (MAD): Number of participants with abnormal findings in 12 Lead Digital electrocardiogram (dECG) | Day 1 to Day 3, Day 5, Day 8 to Day 10
  Safety and tolerability of AZD6793 following oral administration of MAD in healthy participants.
Part 1 (SAD): Number of participants with abnormal findings in Telemetry | Day -1 to Day 3
  Safety and tolerability of AZD6793 following oral administration of SAD in healthy participants.
Part 2 (MAD): Number of participants with abnormal findings in Telemetry | Day -1 to Day 2 and Day 8 to Day 10
  Safety and tolerability of AZD6793 following oral administration of MAD in healthy participants.
Part 1 (SAD): Number of participants with abnormal findings in Physical examinations | From screening, Treatment Day -1 to 4 and follow up visit
  Safety and tolerability of AZD6793 following oral administration of SAD in healthy participants.
Part 2 (MAD): Number of participants with abnormal findings in Physical examinations | From screening, Treatment Day -1 to 10 and follow up visit
  Safety and tolerability of AZD6793 following oral administration of MAD in healthy participants.
Part 1 (SAD): Number of participants with abnormal findings in Laboratory assessments (haematology, serum clinical chemistry, and urinalysis) | From screening, Treatment Day -1, Day 2, Day 4 and Follow up visit (Day 6±1)
  Safety and tolerability of AZD6793 following oral administration of SAD in healthy participants.
Part 2 (MAD): Number of participants with abnormal findings in Laboratory assessments (haematology, serum clinical chemistry, and urinalysis) | From screening, Treatment Day -1 to Day 10 up to Follow up visit (Day 14±1)
  Safety and tolerability of AZD6793 following oral administration of MAD in healthy participants.
Part 3 (Bioavailability): Maximum observed plasma (peak) drug concentration [Cmax] | Day 1 to Day 3
  Evaluating the relative oral bioavailability between the test formulation and the reference formulation after a single oral dose of AZD6793 in healthy participants.
Part 3 (Bioavailability): Area under plasma concentration-time curve from zero to infinity [AUCinf] | Day 1 to Day 3
  Evaluating the relative oral bioavailability between the test formulation and the reference formulation after a single oral dose of AZD6793 in healthy participants.
Part 3 (Food effect): Cmax of AZD6793 | Day 1 to Day 3
  Investigating the effect of a high fat high calorie (HFHC) meal compared to fasting conditions, on the PK of AZD6793 after a single oral dose in healthy participants.
Part 3 (Food effect): AUCinf of AZD6793 | Day 1 to Day 3
  Investigating the effect of a high fat high calorie (HFHC) meal compared to fasting conditions, on the PK of AZD6793 after a single oral dose in healthy participants.
Part 4 (COPD): Number of participants with adverse events | From screening up to Follow up visit (Day 34±2)
  Safety and tolerability of AZD6793 following oral administration repeated up to 28 days (at least 26 days) in COPD participants.
Part 4 (COPD): Number of participants with abnormal findings in vital signs (supine Blood Pressure (BP), pulse, respiratory rate, peripheral oxygen saturation (SpO2) and oral body temperature) | From screening up to Follow up visit (Day 34±2)
  Safety and tolerability of AZD6793 following oral administration repeated up to 28 days (at least 26 days) in COPD participants.
Part 4 (COPD): Number of participants with abnormal findings in 12 Lead electrocardiogram (ECG) | From screening up to Follow up visit (Day 34±2)
  Safety and tolerability of AZD6793 following oral administration repeated up to 28 days (at least 26 days) in COPD participants.
Part 4 (COPD): Number of participants with abnormal findings in Physical examinations | From screening, Treatment Day -1, 1, 14, 28 and follow up visit (34±2)
  Safety and tolerability of AZD6793 following oral administration repeated up to 28 days (at least 26 days) in COPD participants.
Part 4 (COPD): Number of participants with abnormal findings in Laboratory assessments (haematology, clinical chemistry, coagulation tests, and urinalysis) | From screening up to Follow up visit (Day 34±2)
  Safety and tolerability of AZD6793 following oral administration repeated up to 28 days (at least 26 days) in COPD participants.

SECONDARY OUTCOMES:
Part 1 (SAD): Maximum observed plasma (peak) drug concentration (Cmax) | Day 1 to Day 3
  Characterizing pharmacokinetics of AZD6793 following oral administration of SAD in healthy participants.
Part 1 (SAD): Time to reach peak or maximum observed concentration or response following drug administration (tmax) | Day 1 to Day 3
  Characterizing pharmacokinetics of AZD6793 following oral administration of SAD in healthy participants.
Part 1 (SAD): Terminal rate constant, estimated by log linear least squares regression of the terminal part of the concentration time curve (λz) | Day 1 to Day 3
  Characterizing pharmacokinetics of AZD6793 following oral administration of SAD in healthy participants.
Part 1 (SAD): Half life associated with terminal slope (λz) of a semi logarithmic concentration time curve ( t½λz) | Day 1 to Day 3
  Characterizing pharmacokinetics of AZD6793 following oral administration of SAD in healthy participants.
Part 1 (SAD): Partial area under the plasma concentration time curve from time 0 to time 12 (AUC(0-12)) | Day 1 to Day 3
  Characterizing pharmacokinetics of AZD6793 following oral administration of SAD in healthy participants.
Part 1 (SAD): Partial area under the plasma concentration time curve from time 0 to time 24 (AUC(0-24)) | Day 1 to Day 3
  Characterizing pharmacokinetics of AZD6793 following oral administration of SAD in healthy participants.
Part 1 (SAD): Area under the plasma concentration curve from zero to the last quantifiable concentration (AUClast) | Day 1 to Day 3
  Characterizing pharmacokinetics of AZD6793 following oral administration of SAD in healthy participants.
Part 1 (SAD): Area under plasma concentration time curve from zero to infinity (AUCinf) | Day 1 to Day 3
  Characterizing pharmacokinetics of AZD6793 following oral administration of SAD in healthy participants.
Part 1 (SAD): Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | Day 1 to Day 3
  Characterizing pharmacokinetics of AZD6793 following oral administration of SAD in healthy participants.
Part 1 (SAD): Volume of distribution (apparent) at steady state following extravascular administration (based on terminal phase) (Vz/F) | Day 1 to Day 3
  Characterizing pharmacokinetics of AZD6793 following oral administration of SAD in healthy participants.
Part 1 (SAD): Area under the plasma concentration time curve from time zero to time of last quantifiable analyte concentration divided by the dose administered (Dose normalised AUClast) | Day 1 to Day 3
  Characterizing pharmacokinetics of AZD6793 following oral administration of SAD in healthy participants.
Part 1 (SAD): Area under the plasma concentration time curve from time zero extrapolated to infinity divided by the dose administered (Dose normalised AUCinf) | Day 1 to Day 3
  Characterizing pharmacokinetics of AZD6793 following oral administration of SAD in healthy participants.
Part 1 (SAD): Maximum observed plasma (peak) drug concentration divided by the dose administered (Dose normalised Cmax). | Day 1 to Day 3
  Characterizing pharmacokinetics of AZD6793 following oral administration of SAD in healthy participants.
Part 2 (MAD): Maximum observed plasma (peak) drug concentration (Cmax) | Day 1 to Day 10
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 2 (MAD): Concentration at the end of the dosing interval (Ctrough) | Day 1 to Day 10
  Characterizing pharmacokinetics of AZD6793 following oral administration of SAD in healthy participants.
Part 2 (MAD): Temporal change parameter (TCP) assessed in urine | Day 1 and Day 8
  Characterizing pharmacokinetics of AZD6793 following oral administration of SAD in healthy participants.
Part 2 (MAD): Time to reach peak or maximum observed concentration or response following drug administration (tmax) | Day 1 to Day 10
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 2 (MAD): Terminal rate constant, estimated by log linear least squares regression of the terminal part of the concentration time curve (λz) | Day 1 to Day 10
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 2 (MAD): Half life associated with terminal slope (λz) of a semi logarithmic concentration time curve ( t½λz) | Day 1 to Day 10
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 2 (MAD): Partial area under the plasma concentration time curve from time 0 to time 24 (AUC(0-24)) | Day 1 to Day 10
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 2 (MAD): Area under the plasma concentration curve from zero to the last quantifiable concentration (AUClast) | Day 1 to Day 10
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 2 (MAD): Area under plasma concentration time curve from zero to infinity (AUCinf) | Day 1 to Day 10
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 2 (MAD): Area under plasma concentration time curve in the dosing interval t (AUCt) | Day 1 to Day 10
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 2 (MAD): Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | Day 1 to Day 10
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 2 (MAD): Volume of distribution (apparent) at steady state following extravascular administration (based on terminal phase) (Vz/F) | Day 1 to Day 10
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 2 (MAD): Area under the plasma concentration time curve from time zero to time of last quantifiable analyte concentration divided by the dose administered (Dose normalised AUClast) | Day 1 to Day 10
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 2 (MAD): Area under the plasma concentration-time curve from time zero to the dosing interval t concentration divided by the dose administered (Dose normalised AUCt) | Day 1 to Day 10
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 2 (MAD): Maximum observed plasma (peak) drug concentration divided by the dose administered (Dose normalised Cmax) | Day 1 to Day 10
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 2 (MAD): Ratio of the area under the curve (Rac AUC) | Day 1 to Day 10
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 2 (MAD): Accumulation ratio based on Cmax (Rac Cmax) | Day 1 to Day 10
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 2 (MAD): Cumulative amount of unchanged drug excreted into urine from time t1 to time t2 [Ae(t1 t2)] | Day 1 and Day 8
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 2 (MAD): Cumulative amount of unchanged drug excreted into urine (Aeinf) | Day 1 and Day 8
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 2 (MAD): Renal clearance of drug from plasma (CLR) assessed in urine | Day 1 and Day 8
  Characterizing pharmacokinetics of AZD6793 following oral administration of MAD in healthy participants.
Part 3 (Bioavailability): Cmax of AZD6793 (test Vs reference formulation) | Day 1 to Day 3
  To assess the PK profiles of AZD6793 when administered as a test formulation versus reference formulation in healthy participants
Part 3 (Bioavailability): tmax of AZD6793 (test Vs reference formulation) | Day 1 to Day 3
  To assess the PK profiles of AZD6793 when administered as a test formulation versus reference formulation in healthy participants
Part 3 (Bioavailability): λz of AZD6793 (test Vs reference formulation) | Day 1 to Day 3
  To assess the PK profiles of AZD6793 when administered as a test formulation versus reference formulation in healthy participants
Part 3 (Bioavailability): t½λz of AZD6793 (test Vs reference formulation) | Day 1 to Day 3
  To assess the PK profiles of AZD6793 when administered as a test formulation versus reference formulation in healthy participants
Part 3 (Bioavailability): AUC(0-12) of AZD6793 (test Vs reference formulation) | Day 1 to Day 3
  To assess the PK profiles of AZD6793 when administered as a test formulation versus reference formulation in healthy participants
Part 3 (Bioavailability): AUC(0-24) of AZD6793 (test Vs reference formulation) | Day 1 to Day 3
  To assess the PK profiles of AZD6793 when administered as a test formulation versus reference formulation in healthy participants
Part 3 (Bioavailability): AUClast of AZD6793 (test Vs reference formulation) | Day 1 to Day 3
  To assess the PK profiles of AZD6793 when administered as a test formulation versus reference formulation in healthy participants
Part 3 (Bioavailability): AUCinf of AZD6793 (test Vs reference formulation) | Day 1 to Day 3
  To assess the PK profiles of AZD6793 when administered as a test formulation versus reference formulation in healthy participants
Part 3 (Bioavailability): CL/F of AZD6793 (test Vs reference formulation) | Day 1 to Day 3
  To assess the PK profiles of AZD6793 when administered as a test formulation versus reference formulation in healthy participants
Part 3 (Bioavailability): Vz/F of AZD6793 (test Vs reference formulation) | Day 1 to Day 3
  To assess the PK profiles of AZD6793 when administered as a test formulation versus reference formulation in healthy participants
Part 3 (Bioavailability) :Relative bioavailability calculated as test AUC/reference AUC [Frel AUC] | Day 1 to Day 3
  To assess the PK profiles of AZD6793 when administered as a test formulation versus reference formulation in healthy participants
Part 3 (Bioavailability): Relative bioavailability calculated as test Cmax/reference Cmax [Frel Cmax] | Day 1 to Day 3
  To assess the PK profiles of AZD6793 when administered as a test formulation versus reference formulation in healthy participants
Part 3 (Food effect): Cmax of AZD6793 (under fasted and fed state) | Day 1 to Day 3
  To examine the PK profiles of AZD6793 test formulation under fasted and fed (after intake of a HFHC meal) conditions in healthy participants.
Part 3 (Food effect): tmax of AZD6793 (under fasted and fed state) | Day 1 to Day 3
  To examine the PK profiles of AZD6793 test formulation under fasted and fed (after intake of a HFHC meal) conditions in healthy participants.
Part 3 (Food effect): λz of AZD6793 (under fasted and fed state) | Day 1 to Day 3
  To examine the PK profiles of AZD6793 test formulation under fasted and fed (after intake of a HFHC meal) conditions in healthy participants.
Part 3 (Food effect): t½λz of AZD6793 (under fasted and fed state) | Day 1 to Day 3
  To examine the PK profiles of AZD6793 test formulation under fasted and fed (after intake of a HFHC meal) conditions in healthy participants.
Part 3 (Food effect): AUC(0-12) of AZD6793 (under fasted and fed state) | Day 1 to Day 3
  To examine the PK profiles of AZD6793 test formulation under fasted and fed (after intake of a HFHC meal) conditions in healthy participants.
Part 3 (Food effect): AUC(0-24) of AZD6793 (under fasted and fed state) | Day 1 to Day 3
  To examine the PK profiles of AZD6793 test formulation under fasted and fed (after intake of a HFHC meal) conditions in healthy participants.
Part 3 (Food effect): AUClast of AZD6793 (under fasted and fed state) | Day 1 to Day 3
  To examine the PK profiles of AZD6793 test formulation under fasted and fed (after intake of a HFHC meal) conditions in healthy participants.
Part 3 (Food effect): AUCinf of AZD6793 (under fasted and fed state) | Day 1 to Day 3
  To examine the PK profiles of AZD6793 test formulation under fasted and fed (after intake of a HFHC meal) conditions in healthy participants.
Part 3 (Food effect): CL/F of AZD6793 (under fasted and fed state) | Day 1 to Day 3
  To examine the PK profiles of AZD6793 test formulation under fasted and fed (after intake of a HFHC meal) conditions in healthy participants.
Part 3 (Food effect): Vz/F of AZD6793 (under fasted and fed state) | Day 1 to Day 3
  To examine the PK profiles of AZD6793 test formulation under fasted and fed (after intake of a HFHC meal) conditions in healthy participants.
Part 3 (Food effect) :Frel AUC of AZD6793 (under fasted and fed state) | Day 1 to Day 3
  To examine the PK profiles of AZD6793 test formulation under fasted and fed (after intake of a HFHC meal) conditions in healthy participants.
Part 3 (Food effect): Frel Cmax of AZD6793 (under fasted and fed state) | Day 1 to Day 3
  To examine the PK profiles of AZD6793 test formulation under fasted and fed (after intake of a HFHC meal) conditions in healthy participants.
Part 4 (COPD): Maximum observed plasma (peak) drug concentration (Cmax) | Day 1 to Day 28
  Characterizing the pharmacokinetic profile of AZD6793 following oral repeated administration up to 28 days (at least 26 days) in COPD participants
Part 4 (COPD): Concentration at the end of the dosing interval (Ctrough) | Day 1 to Day 28
  Characterizing the pharmacokinetic profile of AZD6793 following oral repeated administration up to 28 days (at least 26 days) in COPD participants
Part 4 (COPD): Temporal change parameter (TCP) assessed in urine | Day 1 and Day 8
  Characterizing the pharmacokinetic profile of AZD6793 following oral repeated administration up to 28 days (at least 26 days) in COPD participants
Part 4 (COPD): Time to reach peak or maximum observed concentration or response following drug administration (tmax) | Day 1 to Day 28
  Characterizing the pharmacokinetic profile of AZD6793 following oral repeated administration up to 28 days (at least 26 days) in COPD participants
Part 4 (COPD): Terminal rate constant, estimated by log linear least squares regression of the terminal part of the concentration time curve (λz) | Day 1 to Day 28
  Characterizing the pharmacokinetic profile of AZD6793 following oral repeated administration up to 28 days (at least 26 days) in COPD participants
Part 4 (COPD): Half life associated with terminal slope (λz) of a semi logarithmic concentration time curve ( t½λz) | Day 1 to Day 28
  Characterizing the pharmacokinetic profile of AZD6793 following oral repeated administration up to 28 days (at least 26 days) in COPD participants
Part 4 (COPD): Partial area under the plasma concentration time curve from time 0 to time 12 (AUC(0-12)) | Day 1 to Day 28
  Characterizing the pharmacokinetic profile of AZD6793 following oral repeated administration up to 28 days (at least 26 days) in COPD participants
Part 4 (COPD): Partial area under the plasma concentration time curve from time 0 to time 24 (AUC(0-24)) | Day 1 to Day 28
  Characterizing the pharmacokinetic profile of AZD6793 following oral repeated administration up to 28 days (at least 26 days) in COPD participants
Part 4 (COPD): Area under the plasma concentration curve from zero to the last quantifiable concentration (AUClast) | Day 1 to Day 28
  Characterizing the pharmacokinetic profile of AZD6793 following oral repeated administration up to 28 days (at least 26 days) in COPD participants
Part 4 (COPD): Area under plasma concentration time curve from zero to infinity (AUCinf) | Day 1 to Day 28
  Characterizing the pharmacokinetic profile of AZD6793 following oral repeated administration up to 28 days (at least 26 days) in COPD participants
Part 4 (COPD): Area under plasma concentration time curve in the dosing interval t (AUCt) | Day 1 to Day 28
  Characterizing the pharmacokinetic profile of AZD6793 following oral repeated administration up to 28 days (at least 26 days) in COPD participants
Part 4 (COPD): Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | Day 1 to Day 28
  Characterizing the pharmacokinetic profile of AZD6793 following oral repeated administration up to 28 days (at least 26 days) in COPD participants
Part 4 (COPD): Volume of distribution (apparent) at steady state following extravascular administration (based on terminal phase) (Vz/F) | Day 1 to Day 28
  Characterizing the pharmacokinetic profile of AZD6793 following oral repeated administration up to 28 days (at least 26 days) in COPD participants
Part 4 (COPD): Ratio of the area under the curve (Rac AUC) | Day 1 to Day 28
  Characterizing the pharmacokinetic profile of AZD6793 following oral repeated administration up to 28 days (at least 26 days) in COPD participants
Part 4 (COPD): Accumulation ratio based on Cmax (Rac Cmax) | Day 1 to Day 28
  Characterizing the pharmacokinetic profile of AZD6793 following oral repeated administration up to 28 days (at least 26 days) in COPD participants

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Research Site, Harrow
  - Research Site, Wythenshawe

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7860C00001&attachmentIdentifier=c63a9d43-3d84-4fed-92c9-dadb3222fe6b&fileName=D7860C00001_Redacted_CSR_Synopsis.pdf&versionIdentifier=